CLINICAL TRIAL: NCT02528487
Title: Predictors of the Long-term Functional Benefits of a Pulmonary Rehabilitation Program?
Status: Suspended | Type: Observational
Why Stopped: Pending financial support
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Collaborators: Mount Sinai Rehabilitation Hospital (Other); Hopital Charles Lemoyne (Other); Centre hospitalier de l'Université de Montréal (CHUM) (Other); Jewish Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Grégory Moullec, Researcher, Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Other Study IDs: 2015-1132 (MP)
Record Dates: First submitted 2015-08-17; First posted 2015-08-19 (Estimated); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Pulmonary Rehabilitation; Chronic Obstructive Pulmonary Disease; Psychiatric Disorders
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Mental Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The present study aims to assess the prevalence and impact of comorbid psychiatric disorders among patients with chronic obstructive pulmonary disease (COPD) undergoing pulmonary rehabilitation (PR), in order to determine the effects of psychiatric comorbidity on exercise tolerance and physical activity post-PR and HRQoL, as well as to determine the processes by which these psychiatric disorders may impact on these patient behaviours.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over the age of 40 will be eligible if
2. they are diagnosed with moderate-severe COPD,
3. currently participate to a PR program, and
4. agree to participate.

Exclusion Criteria:

They will be excluded if:

1. they have any comorbidity that is more important (i.e., more likely to cause morbidity or mortality) than COPD (e.g., active cancer),
2. they have contraindications to exercise (though they will not likely be referred to PR),
3. they have participated in a PR program in the past year,
4. and if they are unable to provide informed consent due to language difficulties or cognitive impairment.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients will be consecutively recruited at entry in one of six PR programs in the Montreal area: Hôpital du Sacré-Coeur de Montréal (HSCM), Mount Sinai Hospital, Hôtel-Dieu de Montréal (CHUM), and Hôpital Charles-LeMoyne, Jewish Rehabilitation Hospital of Laval, McGill University Health Centre (MUHC).
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2015-05 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
The change in exercise tolerance at 1-year post-PR | Participants will be evaluated at 3 time points: (1) post-PR; (2) at 6-mo; (3) at 12-mo follow-up.
  Exercise tolerance will be measured with the 6-minute walking test (6MWT).

SECONDARY OUTCOMES:
The change in health-related quality of life (HRQoL) at 1-year post-PR | Participants will be evaluated at 3 time points: (1) post-PR; (2) at 6-mo; (3) at 12-mo follow-up.
  HRQoL will be measured with the 12-Item Short Form Survey and the COPD Assessment Test

CONTACTS AND LOCATIONS:
Overall Officials: Grégory Moullec, Ph.D., Principal Investigator — Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Locations (5):
- Canada (5):
  - Jewish Rehabilitation Hospital, Laval, Quebec
  - Hopital Charles-Lemoyne, Longueuil, Quebec
  - Hopital du Sacre-Coeur de Montreal, Montreal, Quebec
  - Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - Mount-Sinai Hospital, Montreal, Quebec